CLINICAL TRIAL: NCT07231185
Title: A Phase 2 Open-Label Study to Evaluate the Efficacy, Safety, and Treatment Experience of Hezkue® and Hezkue Turbo® Compared With Select Commercially Available Sildenafil Products in Adult Men With Erectile Dysfunction (ED)
Brief Title: Phase 2 Efficacy Study of Sildenafil Products in Adult Men With Erectile Dysfunction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-011-SIL
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; Viagra; sildenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Hezkue (Experimental): Participants receive Hezkue®, an oral liquid formulation of sildenafil, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Hezkue
- Hezkue Turbo (Experimental): Participants receive Hezkue Turbo®, an oral liquid suspension delivering sildenafil via a metered-dose device, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Hezkue Turbo
- Galotam (Active Comparator): Participants receive Galotam®, a commercially available sildenafil product, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Galotam
- BlueChew (Active Comparator): Participants receive BlueChew® sildenafil chewable tablets, used on an on-demand basis for 12 weeks.
  Interventions: Drug: BlueChew
- Pfizer Viagra (Active Comparator): Participants receive Pfizer Viagra®, a standard oral tablet formulation of sildenafil, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Pfizer Viagra
- Aristo Sildaristo (Active Comparator): Participants receive Aristo Sildaristo®, a commercially available sildenafil tablet product, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Aristo Sildaristo
- Lemonaid Health Viagra (Active Comparator): Participants receive Lemonaid Health-branded sildenafil (Viagra), used on an on-demand basis for 12 weeks.
  Interventions: Drug: Lemonaid Health Sildenafil
- Ro Sparks (Active Comparator): Participants receive Ro Sparks®, a combination sildenafil + tadalafil product, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Ro Sparks
- Hims Hard Mints (Active Comparator): Participants receive Hims Hard Mints®, a combination sildenafil + tadalafil formulation, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Hims Hard Mints
- Hello Cake ED Cake Meds (Active Comparator): Participants receive Hello Cake ED Cake Meds®, a combination sildenafil + tadalafil formulation, used on an on-demand basis for 12 weeks.
  Interventions: Drug: Hello Cake ED Cake Meds

INTERVENTIONS:
Drug: Hezkue — Hezkue® is an oral liquid formulation of sildenafil administered on an on-demand basis for the treatment period.
  Other Names: Sildenafil oral spray
  Arms: Hezkue
Drug: Hezkue Turbo — Hezkue Turbo® is an oral liquid suspension of sildenafil delivered via a metered-dose device, used on an on-demand basis.
  Other Names: Sildenafil liquid suspension
  Arms: Hezkue Turbo
Drug: Galotam — Galotam® is a commercially available sildenafil product administered on an on-demand basis.
  Other Names: Sildenafil tablet (Galotam)
  Arms: Galotam
Drug: BlueChew — BlueChew® sildenafil chewable tablets, used on an on-demand basis.
  Other Names: Sildenafil chewable tablet
  Arms: BlueChew
Drug: Pfizer Viagra — Pfizer Viagra® sildenafil tablets, administered on an on-demand basis.
  Other Names: Sildenafil citrate
  Arms: Pfizer Viagra
Drug: Aristo Sildaristo — Aristo Sildaristo® is a commercially available sildenafil tablet product used on an on-demand basis.
  Other Names: Sildenafil
  Arms: Aristo Sildaristo
Drug: Lemonaid Health Sildenafil — Lemonaid Health-branded sildenafil tablets (Viagra equivalent), administered on an on-demand basis.
  Other Names: Sildenafil (Lemonaid Health)
  Arms: Lemonaid Health Viagra
Drug: Ro Sparks — Ro Sparks® is a combination sildenafil + tadalafil product administered on an on-demand basis.
  Other Names: Sildenafil + Tadalafil (Ro Sparks)
  Arms: Ro Sparks
Drug: Hims Hard Mints — Hims Hard Mints® is a combination formulation containing sildenafil + tadalafil, used on an on-demand basis.
  Other Names: Sildenafil + Tadalafil (Hims)
  Arms: Hims Hard Mints
Drug: Hello Cake ED Cake Meds — Hello Cake ED Cake Meds® is a combination sildenafil + tadalafil product administered on an on-demand basis.
  Other Names: Sildenafil + Tadalafil (Hello Cake)
  Arms: Hello Cake ED Cake Meds

SUMMARY:
The goal of this clinical trial is to learn how different sildenafil-based erectile dysfunction (ED) treatments affect erectile function in adult men. The main questions it aims to answer are:

Does each assigned product improve erectile function over 12 weeks?

What safety or tolerability issues occur when these products are used on an on-demand basis?

Researchers will compare Hezkue® and Hezkue Turbo® with several commercially available sildenafil or sildenafil-plus-tadalafil products to see whether there are differences in effectiveness, treatment experience, or safety.

Participants will:

* Use one assigned ED treatment on demand for 12 weeks
* Complete electronic diaries and questionnaires about sexual-encounter outcomes and treatment satisfaction
* Attend study visits for safety checks, laboratory tests, and assessments of erectile function

DETAILED DESCRIPTION:
This Phase 2, open-label, parallel-group clinical trial evaluates the real-world use of multiple sildenafil-based erectile dysfunction (ED) treatments, including two oral liquid formulations (Hezkue® and Hezkue Turbo®) and several commercially available tablet, chewable, or combination (sildenafil/tadalafil) products. The study is designed to characterize differences in erectile function outcomes, safety profiles, and patient-reported treatment experiences across these products when used on an on-demand basis.

The trial includes a screening period of up to 28 days, followed by 12 weeks of treatment with one assigned product. Participants will use electronic diaries and questionnaires to record sexual-encounter outcomes, timing of effects, treatment satisfaction, and other patient-reported measures. Safety evaluations include adverse event monitoring, vital signs, clinical laboratory assessments, and targeted cardiovascular, ophthalmologic, and otologic examinations.

The design reflects typical on-demand PDE5 inhibitor use and enables comparative assessment across distinct formulations and delivery systems (liquid spray, orodispersible/chewable, and standard tablets). Exploratory analyses will examine work productivity, activity impairment, healthcare utilization, and optional partner-reported measures to better understand the broader impact of ED treatment in daily life.

This description supplements, but does not repeat, information provided in the Brief Summary, Eligibility, or Outcome Measures sections.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18 to 70 years of age.

Documented diagnosis of erectile dysfunction (ED) for at least 3 months, confirmed by a clinician.

Baseline International Index of Erectile Function-Erectile Function (IIEF-EF) domain score ≤25.

Sexually active and attempting sexual intercourse at least 4 times per month during the 3 months prior to screening.

Willing and able to attempt sexual intercourse at least once per week during the study.

Judged by the Investigator to be in good general health other than ED.

Creatinine clearance (CrCl) >80 mL/min as calculated by Cockcroft-Gault.

Able and willing to comply with all study procedures, including use of eDiary/ePRO tools and adherence to dosing instructions.

Exclusion Criteria:

* Use of nitrates or nitric oxide donors in any form.

Use of prohibited antihypertensive medications as defined in the protocol.

Use of phosphodiesterase type 5 (PDE5) inhibitors within 5 days prior to baseline.

Use of CYP450 inhibitors within 14 days prior to first dose.

Use of CYP450 inducers or St. John's Wort within 28 days prior to first dose.

Use of any prescription or non-prescription medications, herbal products, or dietary supplements not approved by the Investigator during the required restriction period.

Known hypersensitivity to sildenafil, tadalafil, vardenafil, peppermint oil, or any component of the investigational product.

Clinically significant abnormalities in screening laboratory tests, vital signs, or electrocardiograms, as judged by the Investigator.

Any hepatic impairment or abnormal liver function test results at screening.

Positive screening test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Clinically significant illness within 30 days prior to the first dose.

Significant cardiovascular disease, including recent myocardial infarction, unstable angina, uncontrolled hypertension, or severe arrhythmias.

History of stroke or neurological disorder that may affect sexual function.

Severe psychiatric disorder or substance abuse that may interfere with study participation.

Anatomical penile deformity (such as Peyronie's disease) that may interfere with erectile function assessments.

Positive urine drug screen for amphetamines, barbiturates, benzodiazepines, cocaine, opiates, phencyclidine (PCP), or MDMA.

Alcohol consumption exceeding 15 units per week.

Initiation of new nicotine products during the study period.

Participation in another clinical trial (other than Hezkue/Hezkue Turbo studies) within 30 days prior to screening.

Blood donation or significant blood loss within 3 months prior to screening, or plasma donation within 14 days prior to screening.

Major surgery within 3 months or minor surgery within 1 month before screening.

Consumption of Seville oranges, grapefruit, or pomelo within 7 days before dosing.

Resting systolic blood pressure outside 90-140 mmHg, diastolic blood pressure outside 50-90 mmHg, or heart rate outside 50-100 beats per minute at screening.

Sexual partner is pregnant or unwilling to use effective contraception during the study.

Any condition that, in the Investigator's opinion, would make the participant unsuitable for the study.

Institutionalized individuals.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in IIEF-EF Domain Score | Baseline to Week 12
  Erectile function will be assessed using the International Index of Erectile Function-Erectile Function (IIEF-EF) domain score, which ranges from 1 to 30, with higher scores indicating better erectile function. Change from baseline to Week 12 will be compared across treatment arms.

SECONDARY OUTCOMES:
SEP-Q2 Penetration Success Rate | Weeks 0-12
  Proportion of "Yes" responses to Sexual Encounter Profile Question 2 (SEP-Q2: ability to achieve vaginal penetration) across all sexual attempts.
SEP-Q3 Intercourse Success Rate | Weeks 0-12
  Proportion of "Yes" responses to Sexual Encounter Profile Question 3 (SEP-Q3: ability to maintain erection through completion of intercourse) across all sexual attempts
Erection Hardness Score (EHS) | Weeks 4, 8, and 12
  Proportion of participants achieving an EHS ≥3 and ≥4 at Weeks 4, 8, and 12.
Global Assessment Question (GAQ) | Week 12
  Proportion of participants responding "Yes" to the GAQ ("Has the treatment improved your erections?").
Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Total Score | Week 12
  Participant-reported satisfaction with erectile dysfunction treatment measured using the EDITS questionnaire.
TSQM-II Scores (Effectiveness, Side Effects, Convenience, Global Satisfaction) | Week 12
  Treatment satisfaction will be assessed using the Treatment Satisfaction Questionnaire for Medication, Version II (TSQM-II). Each TSQM-II domain (Effectiveness, Side Effects, Convenience, and Global Satisfaction) is scored from 0 to 100, with higher scores indicating greater satisfaction in that domain (and fewer perceived side effects on the Side Effects scale).
Time-to-Onset of Effect | Weeks 0-12
  Participant-reported time (in minutes) to erection sufficient for penetration after dosing, recorded via eDiary for each sexual attempt.
Duration of Effect | Weeks 0-12
  Participant-reported duration (in hours) of erectile effect after dosing, recorded via eDiary.
Incidence of Adverse Events (AEs) and Serious AEs (SAEs) | Screening through Week 13
  Frequency and severity of treatment-emergent adverse events, including cardiovascular, ophthalmologic, otologic, and other expected PDE5 inhibitor-related events.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Guralnik, PhD, Study Director — Aspargo Labs, Inc

IPD SHARING:
Plan to Share IPD: No